CLINICAL TRIAL: NCT04521023
Title: A Randomized, Double-blind, Non-inferiority, Multi-center, Phase 4 Trial to Evaluate the Blood Pressure Lowering Effect of a Candesartan/Hydrochlorothiazide(Candemore Plus® Tab) Versus Candesartan/Amlodipine(Cantabell® Tab) in Hypertensive Patients Inadequately Controlled by Candesartan Monotherapy
Brief Title: A Clinical Trial to Evaluate the Blood Pressure Lowering Effect of a Candemore Plus Tab Versus Cantabell Tab in Hypertensive Patients Inadequately Controlled by Candesartan Monotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 244HT16025
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Cantabell Tab
- B (Active Comparator)
  Interventions: Drug: Candemore Plus Tab

INTERVENTIONS:
Drug: Cantabell Tab — Patients assigned to experimental group are treated with Cantabell Tab
  Arms: A
Drug: Candemore Plus Tab — Patients assigned to experimental group are treated with Candemore Plus Tab
  Arms: B

SUMMARY:
Phase 4 clinical trial to Evaluate the blood pressure lowering effect of a Candesartan/Hydrochlorothiazide(Candemore Plus Tab) versus Candesartan/Amlodipine(Cantabell Tab) in Hypertensive Patients

ELIGIBILITY:
Inclusion Criteria:

* over 19 years old
* Agreement with written informed consent
* Hypertensive Patients

Exclusion Criteria:

* Patients with secondary hypertension
* Participated in other trial within 30 days
* In investigator's judgement

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
cSBP(central Systolic Blood Pressure) | change after 8 weeks compared to baseline
  Average cSBP change after 8 weeks compared to baseline

SECONDARY OUTCOMES:
cDBP(central Diastolic Blood Pressure) | change after 8 weeks compared to baseline
  Average cDBP change after 8 weeks compared to baseline
sitSBP(sitting Systolic Blood Pressure) | change after 8 weeks compared to baseline
  Average sitSBP change after 8 weeks compared to baseline
sitDBP(sitting Diastolic Blood Pressure) | change after 8 weeks compared to baseline
  Average sitDBP change after 8 weeks compared to baseline

CONTACTS AND LOCATIONS:
Locations (14):
- South Korea (14):
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Hallym Univ. Medical Center, Anyang
  - Daegu Catholic Univ. Medical Center, Daegu
  - MYONGJI Hospital, Goyang-si
  - Inje University Ilsan Paik Hospital, Ilsan-gu
  - Gachon University Gil Medical Center, Incheon
  - Jeju National University Hospital, Jeju City
  - Gangnam Severance Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - SNU Boramae Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No